CLINICAL TRIAL: NCT06983977
Title: Increasing Physical Activity Among Medical Inpatients by Digital Nudging of Patients and Staff - A Cluster Randomised Multicentre Study
Brief Title: Increasing Physical Activity Among Medical Inpatients by Digital Nudging of Patients and Staff
Acronym: IPAMINA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Christian Dall, Associate professor, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VMK-2403916
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Physical Activity; Inpatients; Digital Health
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Measurement of physical activity
  Interventions: Other: Measurement of physical activity
- Intervention (Experimental): Digital feedback and nudging to participant and staff regarding participants' physical activity levels
  Interventions: Other: Digital nudging

INTERVENTIONS:
Other: Measurement of physical activity — Measurement of physical activity by accelerometer
  Arms: Control
Other: Digital nudging — Digital feedback and nudging to participants (patients) and staff, based on participants' physical activity measurements, aiming to increase patients' physical activity and reduce sedentary time
  Arms: Intervention

SUMMARY:
Sedentary behaviour among medical inpatients is strongly associated with hospital-associated functional decline and poses a severe threat to patients' functional capacity and independency. High human and socioeconomic costs underline the urgency to find solutions to this world-wide problem.

Objective: This multicentre study, including a total of 400 patients from Copenhagen, Aalborg, Tórshavn, and Nuuk, will assess the effect of a digital intervention that aims to reduce sedentary behaviour and increase physical activity in medical inpatients.

Intervention: Digital feedback and nudging regarding the patients' physical activity levels to patients and healthcare staff Design: Stepped-wedge cluster randomised multicentre trial Primary outcome: Daily average time of patients' physical activity (minutes).

ELIGIBILITY:
Inclusion Criteria:

* Admitted to one of the participating wards
* Has understood and signed informed consent
* Reads and understands Danish, Faroese, Greenlandic or English

Exclusion Criteria:

* Has an expected hospitalisation less than 24 hours after potential recruitment
* Is not able to give informed consent to participate in the study
* Has allergy towards band aid
* Not able to (shortly) stand in an upright position even with maximal assistance
* There are contraindications for the patient to mobilise or be physically active due to unstabilized acute medical conditions, including, but not limited to, acute aortic dissection, -myocardial infarction, -pulmonary embolism, -sepsis.
* There are ethical concerns regarding the patients' participation in the study, including, but not limited to, the patient being:

  * In the terminal phase of life
  * In a crisis state regarding their disease/situation and deemed unfit for participation

To ensure medically responsible inclusion of patients, the project personnel will consult and confer with the treatment responsible medical doctor, or their delegate, before including a potential participant for the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Daily average time of participants' physical activity (minutes) | From enrollment to end of trial participation (maximum 7 days)

CONTACTS AND LOCATIONS:
Overall Officials: Christian H Dall, Associate professor, PhD, Principal Investigator — Bispebjerg Hospital
Locations (4):
- Denmark (2):
  - Bispebjerg Hospital, Copenhagen, Capital Region
  - Aalborg University Hospital, Hobro, North Denmark
- National Hospital, Tórshavn, Faroe Islands
- Queen Ingrids Hospital, Nuuk, Greenland

IPD SHARING:
Plan to Share IPD: No